CLINICAL TRIAL: NCT00977730
Title: The Effect of the Dietary Supplement Protandim on Non-Alcoholic Steatohepatitis: A Randomized, Double Blind, Placebo-Controlled Study
Brief Title: The Effect of Protandim on Non-alcoholic Steatohepatitis
Acronym: NASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-0848
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2009-09

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: Hepatitis; Fatty Liver; Non Alcoholic Steatohepatitis; Protandim
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis; Fatty Liver | interventions — Protandim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protandim (Active Comparator)
  Interventions: Dietary Supplement: Protandim
- Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Protandim — 1 675 mg capsule Protandim PO/day vs. 1 sugar pill PO/day
  Arms: Protandim
Dietary Supplement: Placebo — 1 675 mg capsule Protandim PO/day vs. 1 sugar pill PO/day
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to evaluate the effect of Protandim on the degree of liver injury after one year of supplementation. Protandim is a nutritional supplement composed of the following 5 botanical extracts: Bacopa Moniera extract, Milk Thistle extract, Ashwagandha powder, Green tea, and Turmeric extract. Protandim is commercially available and can be purchased without a prescription. Our findings could lead to a better understanding of the role of oxidative stress and antioxidant therapy in NASH and may ultimately help improve patient care.

Hypothesis #1: Protandim will lead to a significant improvement in NAS compared to placebo.

Hypothesis #2: Protandim will lead to a significant decrease in serum markers of oxidative stress and liver chemistry tests.

Hypothesis #3: Protandim will lead to decreased levels of TNF- α compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry at least 18 years.
* Serum alanine (ALT) aminotransferase activity that is above the upper limits of normal.
* Evidence of steatohepatitis on liver biopsy performed within the previous 6 months with a NAFLD activity score (NAS) of at least 3 (of a total possible score of 8) including a score of at least 1 each for steatosis, hepatocellular injury and parenchymal inflammation. Histological criteria of steatohepatitis include: (1) macrovesicular steatosis, (2) acinar zone 3 hepatocellular injury (ballooning degeneration), (3) parenchymal inflammation, and (4) portal inflammation. Additional (but not required) features include the presence of (5) Mallory's hyaline and (6) pericellular and/or sinusoidal fibrosis that predominantly involves zone 3.
* Written informed consent.
* Willingness to have a repeat percutaneous liver biopsy following 1 year of supplementation.

Exclusion Criteria:

* Evidence of another form of liver disease as evidenced by any of the following:

  1. Hepatitis B, as defined by the presence of hepatitis B surface antigen (HBsAg).
  2. Hepatitis C, as defined by the presence of hepatitis C virus (HCV) antibody or HCV RNA in serum.
  3. Autoimmune hepatitis, as defined by anti-nuclear antibody (ANA) of 1:160 or greater (or positive smooth muscle antibody) and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
  4. Autoimmune cholestatic liver disorders, as defined by elevation of anti-mitochondrial antibody of greater than 1:80 (or positive AMA by lab report if a titer is not given) or liver histology consistent with primary biliary cirrhosis or primary (or secondary) sclerosing cholangitis.
  5. Wilson's disease, as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson's disease.
  6. Alpha-1-antitrypsin deficiency, as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
  7. Iron overload/hemochromatosis, as defined by the following: elevated transferrin saturation (greater than 45 percent) OR serum ferritin (> 300 microg/L in men or >200 microg/L in women), with one of the following: 1) presence of 3+ or 4+ stainable iron on liver biopsy (if obtained); or 2) Hemochromatosis gene testing showing homozygosity for C282Y or compound heterozygosity for C282Y/H63D (if obtained).
  8. Drug-induced liver disease, as defined on the basis of typical exposure and history.
  9. Intrahepatic and/or extrahepatic duct obstruction, as shown by imaging studies (if obtained).
* History of excess alcohol ingestion, averaging more than 40 gm/day (3 drinks per day) at any time in the previous 10 years, or history of alcohol intake averaging greater than 40 gm/week (3 drinks/week) in the previous year.
* Contraindications to liver biopsy: platelet counts less than 75,000/mm(3) or INR>1.4.
* Stage III or IV fibrosis on baseline liver biopsy.
* History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis including (but not limited to) corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.
* Presence of diabetes mellitus as defined by any of the following: 1) fasting plasma glucose of greater than or equal to 126 mg/dl on 2 separate occasions; or 2) diabetic symptoms with a history of random plasma glucose of greater than or equal to 200 mg/dl.
* Use of anti-diabetic drugs, including insulin, biguanides, sulfonylureas, weight loss medications (either over the counter or prescription), or thiazolidinediones in the previous 6 months. Use of these medications will also be prohibited for the duration of the study.
* Use of cholesterol lowering medications, including statins.
* Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease with hypoxia, renal failure, organ transplantation, serious psychiatric disease, HIV, or malignancy that, in the opinion of the investigator would preclude adequate follow up.
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.
* Pregnancy.
* Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study that is suggestive of liver cancer.
* Serum creatinine greater than 1.5 mg/dl in men and greater than 1.3 mg/dl in women.
* Body habitus or other patient issues that necessitated the original liver biopsy being obtained through radiology (by transjugular approach).
* Abnormal thyroid function, as indicated by an abnormal screening TSH.
* Total Bilirubin > 2.0
* AST or ALT > 3 times the upper limits of normal.
* Serum Sodium <130
* Hematocrit < 35
* Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study.
* Use of any herbal or non-prescription medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in NAS at study completion in the Protandim group compared to the placebo group. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Austin, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Denver, Colorado, United States